CLINICAL TRIAL: NCT00859482
Title: A Phase IV Study to Investigate Differential Immune Effects of Natalizumab
Brief Title: Differential Immune Effects of Natalizumab
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Norman Putzki, MD, Cantonal Hospital St. Gallen
Other Study IDs: Ntz-Tregs1
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Sclerosis, Relapsing Remitting
Keywords: natalizumab; multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — full blodd
Oversight: Data Monitoring Committee: No

SUMMARY:
Natalizumab is a humanized monoclonal antibody directed against Very Late Activation Antigene 4 (VLA-4) and has a potent effect on disease activity in multiple sclerosis (MS). A blockade of VLA-4 with natalizumab may not only interfere with autoimmunological processes but also with central nervous system (CNS) immune surveillance.

DETAILED DESCRIPTION:
Longitudinal ex vivo and in vitro study to determine the effect of natalizumab on frequency of distinct immune cells and on the frequency and suppressive function of natural CD4+CD25+ regulatory T cells (Tregs).

ELIGIBILITY:
Inclusion Criteria:

* relapsing remitting MS
* indication for natalizumab treatment

Exclusion Criteria:

* other disease modifying agents within 2 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initiating natalizumab for treatment of relapsing remitting MS
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Function of T regulatory cells | at month 3

SECONDARY OUTCOMES:
Change in distinct immune cell lines | month 3

CONTACTS AND LOCATIONS:
Overall Officials: Norman Putzki, MD, Principal Investigator — KSSG, 9007 St. Gallen, Switzerland